CLINICAL TRIAL: NCT05649176
Title: Lifestyle Intervention for Improving Metabolic and Motivational Outcomes
Brief Title: Lifestyle Intervention for Improving Insulin Resistance and Concern for Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Candida Rebello, Assistant Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PBRC 2022-028; 4R00AG065419-03 (NIH)
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Insulin Sensitivity; Apathy
MeSH Terms: conditions — Insulin Resistance; Lethargy | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Randomized controlled two-arm parallel trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a feeding study. All participants will receive a diet designed to moderate the blood glucose response. The diets will be similar except that in the experimental group soybean flour (soy) will be incorporated into the foods
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet without soy (Active Comparator): Participants receive a diet to moderate the blood glucose response that does not include soy
  Interventions: Other: Diet without soy
- Diet with soy (Experimental): Participants receive a diet to moderate the blood glucose response that includes soy
  Interventions: Other: Diet with soy

INTERVENTIONS:
Other: Diet without soy — The diet is designed to moderate the blood glucose response with a similar macronutrient composition as the experimental diet but does not contain soy.
  Other Names: Low glycemic index and reduced energy density
  Arms: Diet without soy
Other: Diet with soy — The diet is designed to moderate the blood glucose response with a similar macronutrient composition as the comparator diet but contains soy.
  Other Names: Low glycemic index and reduced energy density
  Arms: Diet with soy

SUMMARY:
The primary objective of this study is to test the effect of a diet and exercise program in older adults with insulin resistance and a motivation disorder known as apathy. The main questions the study aims to answer are:

1. Does the diet and exercise program improve insulin resistance and apathy?
2. Does the addition of soybean to the diet enhance the effect? Participants will be given all meals for 12 weeks and will exercise under supervision. They will undergo a test of insulin sensitivity and complete questionnaires.

Researchers will compare the groups given:

1. A diet to moderate the blood glucose response that contains soybean; and
2. A diet to moderate the blood glucose response that does not contain soybean.

DETAILED DESCRIPTION:
This randomized trial will examine the blood glucose moderating effect of a diet and exercise program in 40 older adults with obesity, insulin resistance, and apathy. The primary objective of this study is to examine the effect of a diet and exercise program on insulin sensitivity and apathy and determine if the addition of soybean to the diet enhances the effect. The primary outcomes of the study are insulin sensitivity measured using the hyperinsulinemic euglycemic clamp test and apathy evaluated using the Apathy Evaluation Scale.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) greater than or equal to 30kg/m2
* Mini-Mental State Examination (MMSE) > 25
* Geriatric Depression Scale-15 (GDS-15) < 6
* Apathy Evaluation Scale - score > 30 or GDS-15 Apathy subscale - score ≥ 2
* Homeostatic model assessment of insulin resistance (HOMA-IR) ≥ 3
* Sedentary: < 90 minutes of moderate to vigorous physical activity/week.

Exclusion Criteria:

* Subjects with a diagnosis of Type 2 diabetes received more than five years ago.
* Participants who have type 1 diabetes
* Participants being treated with prescription or over the counter medications that have a significant effect on insulin resistance, obesity, high density lipoprotein cholesterol, triglycerides, metabolic rate and those that significantly increase body weight.
* Participants who are on concomitant therapy with glucocorticoids.
* Participants with evidence and/or history (within the preceding 6 months) of significant gastrointestinal dysfunction.
* Participants that have had a fluctuation in body weight >5% in the preceding 2 months.
* Any other conditions that may impede testing of the study hypothesis.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 12 weeks
  Insulin sensitivity will measured in a hyperinsulinemic euglycemic clamp test
Apathy | 12 weeks
  Apathy will be evaluated using the Apathy Evaluation Scale

CONTACTS AND LOCATIONS:
Overall Officials: Candida J Rebello, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Solomon TP, Haus JM, Kelly KR, Cook MD, Filion J, Rocco M, Kashyap SR, Watanabe RM, Barkoukis H, Kirwan JP. A low-glycemic index diet combined with exercise reduces insulin resistance, postprandial hyperinsulinemia, and glucose-dependent insulinotropic polypeptide responses in obese, prediabetic humans. Am J Clin Nutr. 2010 Dec;92(6):1359-68. doi: 10.3945/ajcn.2010.29771. Epub 2010 Oct 27. PMID 20980494
- [Background] Solomon TP, Haus JM, Kelly KR, Cook MD, Riccardi M, Rocco M, Kashyap SR, Barkoukis H, Kirwan JP. Randomized trial on the effects of a 7-d low-glycemic diet and exercise intervention on insulin resistance in older obese humans. Am J Clin Nutr. 2009 Nov;90(5):1222-9. doi: 10.3945/ajcn.2009.28293. Epub 2009 Sep 30. PMID 19793849